CLINICAL TRIAL: NCT07403162
Title: Effects of Cuevas Medek Exercises on Postural Control and Balance in Children With Spastic Cerebral Palsy
Brief Title: Cuevas Medek Exercises to Improve Postural Control and Balance in Children With Spastic Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02330 Rimsha Waheed
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Spastic Cerebral Palsy (sCP)
Keywords: Cerebral palsy; Postural balance; Postural control; Pediatric physical therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Masking Description: This is an open-label study as blinding of participants and therapists is not feasible due to the nature of the physiotherapy interventions. Outcome assessments will be conducted using standardized assessment tools to reduce assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cuevas medek exercise (Experimental): Children in this group will receive Cuevas Medek Exercises focusing on activation of postural responses and balance control through progressively challenging activities during the intervention period
  Interventions: Other: Cuevas medek exercises
- Conventional therapy (Active Comparator): Children in this group will receive conventional physiotherapy including stretching, strengthening, and task-oriented activities aimed at improving postural control and balance
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Other: Cuevas medek exercises — Children will receive Cuevas Medek Exercises 3 sessions per week, at an appropriate effort level guided by the therapist, each session lasting 30 minutes, focusing on dynamic postural activation, balance reactions, and functional movement tasks
  Other Names: CME
  Arms: cuevas medek exercise
Other: Conventional Therapy — Children will receive conventional physiotherapy 3 sessions per week, at moderate effort suitable for age and condition, each session 30 minutes long, including stretching, strengthening, and task-oriented activities to improve postural control and balance
  Arms: Conventional therapy

SUMMARY:
This study aims to evaluate the effects of Cuevas Medek Exercises on postural control and balance in children with spastic cerebral palsy. Children meeting the eligibility criteria will be randomly allocated into two groups receiving Cuevas Medek Exercises or conventional therapy. The outcomes will be assessed before and after the intervention period to determine the effectiveness of the intervention.

DETAILED DESCRIPTION:
Spastic cerebral palsy is a common condition characterized by impaired postural control, poor balance, and limitations in functional movement, which affect a child's ability to maintain stability during daily activities. Conventional physiotherapy is commonly used to address these impairments through strengthening, stretching, and task-based exercises, with variable functional outcomes.

Cuevas Medek Exercises is a dynamic therapeutic approach that focuses on activating automatic postural responses and balance reactions through progressively challenging activities with minimal external support. While this approach has shown potential benefits in improving motor control and postural responses, evidence comparing its effects on postural control and balance with conventional therapy in children with spastic cerebral palsy remains limited.

Therefore, a randomized controlled trial is needed to compare the effects of Cuevas Medek Exercises and conventional therapy on postural control and balance in children with spastic cerebral palsy, with the aim of providing evidence to support clinical decision-making in pediatric physiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with spastic diplegic cerebral palsy
* GMFCS Level III to V
* Modified Ashworth Scale ≤ 2
* Able to follow simple commands

Exclusion Criteria:

* Severe cognitive impairment
* Uncontrolled epilepsy or frequent seizures
* Visual or hearing impairment limiting treatment
* History of recent orthopedic or neurosurgical procedures
* Other neurological disorders (genetic syndromes, traumatic brain injury)
* Participation in other experimental therapies during the study period

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Postural Control | At the end of 4 weeks of intervention
  Changes from baseline in postural control will be assessed using the Posture and Postural Ability Scale (PPAS). The scale evaluates the child's ability to maintain posture during functional tasks and measures automatic postural responses. The PPAS consists of several domains including trunk control, limb alignment, and dynamic balance. The scoring ranges from 0 to 30, where 0 indicates no disability and 30 indicates maximum postural impairment.

SECONDARY OUTCOMES:
Balance | At the end of 4 weeks of intervention
  Changes from baseline in balance will be assessed using the Pediatric Balance Scale (PBS). The PBS evaluates balance in sitting, standing, and during functional tasks such as reaching and turning. The scale consists of 14 items, each scored from 0 to 4, giving a total score ranging from 0 (poor balance) to 56 (excellent balance).

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Bashir, PhD, Principal Investigator — Riphah International University
Locations (1):
- Tehsil Headquarter Bhalwal, Bhalwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferreira AD, Gerzson LR, de Almeida CS, Lopes GB. Cuevas Medek exercises a neurological rehabilitation for children, the effect in developmental hip dysplasia in a patient with cerebral palsy: case study. Arquivos de Neuro-Psiquiatria. 2023;81(S 01):A056.
- [Background] Mitroi S. Stimulation of triple extension tone and orthostatic balance in the child with cerebral palsy through exercises specific to Medek method. Physical Education, Sport and Kinesiology Journal. 2016;1(43):48-51
- [Background] Milne N, Neustaeter A, Thomas H, Ritter M, Macdonald K. Review Protocol: EXPLORING THE EFFECTIVENESS OF CUEVAS MEDEK EXERCISES (CME) IN PAEDIATRIC POPULATIONS: A SYSTEMATIC SCOPING REVIEW. 2023
- [Background] Yun G, Huang M, Cao J, Hu X. Selective motor control correlates with gross motor ability, functional balance and gait performance in ambulant children with bilateral spastic cerebral palsy. Gait & posture. 2023;99:9-13
- [Background] Adıguzel H, Elbasan B. Effects of modified pilates on trunk, postural control, gait and balance in children with cerebral palsy: a single-blinded randomized controlled study. Acta Neurologica Belgica. 2022;122(4):903-14
- [Background] Elnaggar RK, Ramirez-Campillo R, Azab AR, Alrawaili SM, Alghadier M, Alotaibi MA, et al. Optimization of postural control, balance, and mobility in children with cerebral palsy: A randomized comparative analysis of independent and integrated effects of Pilates and Plyometrics. Children. 2024;11(2):243
- [Background] Crenshaw JR, Petersen DA, Conner BC, Tracy JB, Pigman J, Wright HG, et al. Anteroposterior balance reactions in children with spastic cerebral palsy. Developmental Medicine & Child Neurology. 2020;62(6):700-8
- [Background] Bickley C, Linton J, Sullivan E, Mitchell K, Slota G, Barnes D. Comparison of simultaneous static standing balance data on a pressure mat and force plate in typical children and in children with cerebral palsy. Gait & posture. 2019;67:91-8.
- [Background] Woollacott MH, Shumway-Cook A. Postural dysfunction during standing and walking in children with cerebral palsy: what are the underlying problems and what new therapies might improve balance? Neural Plast. 2005;12(2-3):211-9; discussion 263-72. doi: 10.1155/NP.2005.211. PMID 16097489
- [Background] Paul S, Nahar A, Bhagawati M, Kunwar AJ. A review on recent advances of cerebral palsy. Oxidative medicine and cellular longevity. 2022;2022(1):2622310.
- [Background] Gulati S, Sondhi V. Cerebral palsy: an overview. The Indian Journal of Pediatrics. 2018;85:1006-16.
- [Background] Novak I, McIntyre S, Morgan C, Campbell L, Dark L, Morton N, Stumbles E, Wilson SA, Goldsmith S. A systematic review of interventions for children with cerebral palsy: state of the evidence. Dev Med Child Neurol. 2013 Oct;55(10):885-910. doi: 10.1111/dmcn.12246. Epub 2013 Aug 21. PMID 23962350